CLINICAL TRIAL: NCT02489084
Title: Predictive Models for Radiation-induced Side Effects in Head and Neck Cancer Based on Single Nucleotide Polymorphisms (SNP)
Acronym: HANS
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: RT2011-03
Record Dates: First submitted 2015-05-19; First posted 2015-07-02 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck neoplasms; Genome-wide association study; Polymorphism, single nucleotide; Toxicity
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood sampling

SUMMARY:
Background of the study:

Swallowing dysfunction and xerostomia are the most frequently reported radiation-induced side effects (RISE) after (chemo) radiation ((CH) RT) in head and neck cancer (HNC) patients and have a major impact on the general dimensions of quality of life (QoL). In radiation0oncology, normal tissue complication probability (NTCP) models based on dose-volume parameters being used to determine the risk of acute and late RISE. NTCP models containing genetic determinants of radiosensitivity, such as single nucleotide polymorphisms (SNPs), may improve model performance and thus enable more individualized radiotherapy. Information of the predictive value of SNPs or SNP signatures among patients with HNC is currently not available.

Objective of the study:

The main objective of this project will be to test the hypothesis that SNP profiles can improve the performance of predictive models for the most frequently reported late RISE, i.e. dysphagia, in HNC patients after curative (CH) RT. Secondary objectives will be improvement of NTCP models for HNC patients by adding SNP profiles predictive of (1) acute mucositis; (2) acute dysphagia; (3) salivary dysfunction; (4) acute xerostomia; (5) late xerostomia; (6) osteoradionecrosis; (7) hypothyroidism; (8) patient-rated HNC symptoms and ; (9) quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven head and neck cancer
* Primary site in the oral cavity, oropharynx, hypopharynx, nasopharynx, paranasal sinuses, and/or salivary glands
* Treatment with curative intent with primary or postoperative radiotherapy either or not combined with systemic treatment
* Northern European ethnicity (ethnicity is a known confounder in SNP association studies)
* Willing and able to comply with the study prescriptions
* 18 years or older
* No prior radiation (in the head and neck area)
* Patients must have sufficient knowledge of the Dutch language to understand the meaning of the study as described in the patient information
* Have given written informed consent before patient registration

Exclusion Criteria:

* Prior radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients ≥18 years still alive and treated since April 2007 for HNC at the department of Radiation Oncology of the UMCG, Groningen, the Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-09; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in acute toxicity | At 1,2,3,4,5,6,7 and 12 weeks after first day of radiation therapy
  Dysphagia; mucositis; salivary dysfunction; xerostomia
Change in late toxicity | At 6,12,18,24,36,48,60 months after last day of completion of treatment
  Dysphagia; xerostomia; osteoradionecrosis; hypothyroidism
Change in patient-rated symptoms | At 1,2,3,4,5,6,7 and 12 weeks after first day of radiation therapy
  Assessed by questionnaires
Change in patient-rated Quality-of-Life | At 6,12,18,24,36,48,60 months after last day of completion of treatment
  Assessed by questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands